CLINICAL TRIAL: NCT04155645
Title: A Phase I Randomized, Single-blind, Placebo-controlled Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of AZD8233 Following Multiple Ascending Subcutaneous Dose Administration in Subjects With Dyslipidemia With or Without Type 2 Diabetes
Brief Title: To Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of AZD8233 After Multiple Dose Administration in Subjects With Dyslipidemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D7990C00002
Record Dates: First submitted 2019-11-05; First posted 2019-11-07 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: Dyslipidemia
Keywords: Multiple Ascending Dose; AZD8233; Safety; Tolerability; PK; PD
MeSH Terms: conditions — Dyslipidemias

STUDY DESIGN:
Who Masked: Participant
Masking Description: This study is single-blind with regards to treatment (AZD8233 or placebo) at each dose level. AZD8233 and placebo will be matched for appearance and amount. Subjects randomized to placebo will receive the same volume of injection as subjects on active drug.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cohort 1 (Experimental): On Days 1, 8, 29, and 57, randomized subjects will receive SC dose of AZD8233 dose 1 injection (8 subjects) or matching placebo (3 subjects).
  Interventions: Drug: AZD8233 subcutaneous injection; Drug: Placebo
- Cohort 2 (Experimental): On Days 1, 8, 29, and 57, randomized subjects will receive SC dose of AZD8233 dose 2 injection (8 subjects) or matching placebo (3 subjects).
  Interventions: Drug: AZD8233 subcutaneous injection; Drug: Placebo
- Cohort 3 (Experimental): On Days 1, 8, 29, and 57, randomized subjects will receive SC dose of AZD8233 dose 3 injection (8 subjects) or matching placebo (3 subjects).
  Interventions: Drug: AZD8233 subcutaneous injection; Drug: Placebo

INTERVENTIONS:
Drug: AZD8233 subcutaneous injection — Randomized subjects will receive SC dose of AZD8233 (dose 1, dose 2, and dose 3) injection.
Drug: Placebo — Randomized subjects will receive SC dose of placebo injection.

SUMMARY:
This is a Phase I study to assess the safety, tolerability and pharmacokinetics (PK), and pharmacodynamics (PD) of AZD8233, following subcutaneous (SC) administration of multiple ascending doses (MAD) of AZD8233 in subjects with confirmed dyslipidemia with or without type 2 diabetes.

DETAILED DESCRIPTION:
This study is a Phase 1, randomized, single-blind, placebo-controlled, multiple dose group design in up to 33 male or female subjects with dyslipidemia with or without Type 2 diabetes and performed at multiple study centers. The planned number of cohorts is 3 but up to 5 cohorts may be included if the Safety Review Committee (SRC) considers it necessary. The 3 multiple dose levels of SC AZD8233 planned are:

* Cohort 1: Dose 1 (starting dose).
* Cohort 2: Dose 2 (provisional dose).
* Cohort 3: Dose 3 (provisional dose). Within each of these cohorts, 8 subjects will be randomized to receive AZD8233 and 3 subjects randomized to receive placebo. Cohorts 2 and 3 may be run in parallel if Cohort 3 is a lower dose. If Cohort 3 is a higher dose, the cohorts will be run sequentially. At any time, the dose levels may be adapted by the SRC based on emerging data. The expected duration of each patient in this study is up to 28 weeks with a maximum of 17 visits. Screening will be completed between Days -28 and -1. Each subject will receive single doses of AZD8233 or placebo on Days 1, 8, 29, and 57. The treatment period will consist of 58 days (up to Visit 9), followed by a follow-up period (up to Visit 17).

Following review of data, the SRC may decide to adjust the following for subsequent cohorts:

* The timing and amount of the loading dose.
* The length of the stay at the study site, the timing and number of assessments and/or samples.
* As decided by the SRC, blood and urine samples collected in the study may be used to address any of the other pre-specified study objectives.
* Each subject will be followed up for 16 weeks post last dose.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated, written informed consent before any study specific procedures.
2. Must be willing and able to comply with all required study procedures.
3. Male or female subjects aged 18 to 65 years at signing of informed consent.
4. Females must not be pregnant and must have a negative urine pregnancy test at the Screening Visit and on admission to the Clinical Unit, must not be lactating; or must be of non-childbearing potential, confirmed at the Screening Visit by fulfilling one of the following criteria:

   * Postmenopausal defined as 12 months with no menses without an alternative medical cause.
   * Documentation of irreversible surgical sterilization by hysterectomy, bilateral oophorectomy, or bilateral salpingectomy but not tubal ligation.
5. Have suitable veins for cannulation or repeated venipuncture.
6. Have a body mass index between 25 and 40 kg/m2.
7. Have a Low-density lipoprotein (LDL) cholesterol > 70 but <190 mg/dL (4.9 mmol/L).
8. Calculated glomerular filtration rate > 60 mL/min by estimated glomerular filtration rate using chronic kidney disease epidemiology equations.
9. Subjects should be receiving moderate- or high-intensity statin therapy as defined by the American College of Cardiology/American Heart Association guideline on blood cholesterol management
10. Subjects should be on stable medication for a certain time period prior to randomization.
11. Provision of signed, written, and dated informed consent for mandatory and optional genetic research. All subjects in the study, except for healthy volunteers, need to consent to the mandatory genetic component of the study and sign the consent form for the main study.
12. If a healthy volunteer population is included by the SRC, then screen for eligibility criteria and study restrictions for healthy volunteer population.

Exclusion criteria:

1. History or presence of gastrointestinal, hepatic or renal disease or any other condition known to interfere with absorption, distribution, metabolism or excretion of drugs.
2. Any uncontrolled or serious disease, or any medical (known major active infection or major hematological, renal, metabolic, gastrointestinal or endocrine dysfunction) or surgical condition that, in the opinion of the Investigator, may either interfere with participation in the clinical study and/or put the participant at significant risk.
3. Blood dyscrasias with increased risk of bleeding including idiopathic thrombocytopenic purpura and thrombotic thrombocytopenic purpura or symptoms of increased risk of bleeding (frequent bleeding gums or nose bleeds).
4. History of major bleed or high-risk of bleeding diathesis.
5. Subjects ≥ 20 years of age with a high 10-year risk of heart disease or stroke as calculated using the atherosclerotic cardiovascular disease (ASCVD) Risk Estimator.
6. Malignancy (except non-melanoma skin cancers, cervical in-situ carcinoma, breast ductal carcinoma in-situ, or Stage 1 prostate carcinoma) within the last 10 years.
7. Recipient of any major organ transplant, eg, lung, liver, heart, bone marrow, renal.
8. LDL or plasma apheresis within 12 months prior to randomization.
9. Uncontrolled hypertension defined as supine SBP >160 mmHg or DBP >90 mmHg.
10. Heart rate after 10 minutes supine rest <50 or >100 bpm.
11. Any laboratory values with the following deviations at the Screening Visit or Day -1, test may be repeated at the discretion of the Investigator if abnormal: Any positive result on screening for serum hepatitis B surface antigen, hepatitis C antibody, and human immunodeficiency virus; ALT > 1.5 times (Upper limit of normal [ULN]); AST >1.5 times ULN; Creatinine > 1.5 mg/dL; WBC < lower limit of normal (LLN); Hemoglobin < 12 g/dL in men or < 11 g/dL in women; Platelet count ≤ LLN; activated partial thromboplastin time > ULN and prothrombin time > ULN; urinary albumin-to-creatinine ratio > 11 mg/μmol.
12. Any clinically important abnormalities in rhythm, conduction or morphology of the resting ECG and any clinically important abnormalities in the 12-lead ECG as considered by the Investigator that may interfere with the interpretation of QTc interval (QTcF > 450 ms) changes, including abnormal ST-T-wave morphology, particularly in the protocol defined primary lead or left ventricular hypertrophy, test may be repeated at the discretion of the Investigator if abnormal.
13. Males who are unwilling to use an acceptable method of birth control during the entire study period. Acceptable methods of preventing pregnancy are true abstinence or use together, with their female partner/spouse, birth control pills, injections, implants, patches, or intrauterine devices in combination with a barrier method. A barrier method is not necessary if the female partner is sterilized.
14. Known or suspected history of drug abuse by the Investigator. 15, Smokers with > 10 cigarettes/day and unable to comply with the nicotine restriction during the study.

16. History of alcohol abuse or excessive intake of alcohol as judged by the Investigator.

17. Positive screen for drugs of abuse at the Screening Visit or admission to the study site.

18. Excessive intake of caffeine-containing drinks or food (eg, coffee, tea, chocolate,) as judged by the Investigator.

19. Use of drugs with cytochrome 450 enzyme inducing properties such as St John's Wort within 3 weeks before the first administration of investigational medicinal product (IMP).

20. Insulin or glucagon-like peptide 1 receptor agonist therapy during last 3 months prior to randomization.

21. Anti-platelet therapy, other than low dose aspirin ≤ 100 mg/day, within 1 month prior to randomization.

22. Mipomersen, or lomitapide within 12 months prior to randomization. 23. Proprotein convertase subtilisin/kexin type 9 inhibition treatment within 6 months prior to randomization.

24. Use of any herbal remedies, megadose vitamins (intake of 20 to 600 times the recommended daily dose) and minerals during the 2 weeks prior to the first administration of IMP or 5 half-lives, whichever is longer.

25. Previous administration of AZD8233/AZD6615. 26. Received another new chemical entity within 30 days of last follow-up to first administration of the IMP of this study or 5 half-lives from last dose to first administration of IMP, whichever is the longest.

27. Plasma donation within 1 month of the Screening Visit or any blood donation/blood loss > 500 mL during the 3 months before the Screening Visit.

28. History of severe allergy/hypersensitivity or ongoing clinically important allergy/hypersensitivity, as judged by the Investigator or history of hypersensitivity to drugs with a similar chemical structure or class to AZD8233.

29. Involvement of any Astra Zeneca or study site employee or their close relatives.

30. Subjects who cannot communicate reliably with the Investigator. 31. Vulnerable subjects, eg, kept in detention, protected adults under guardianship, trusteeship, or committed to an institution by governmental or juridical order.

32. Any clinically important illness, medical/surgical procedure or trauma within 4 weeks of the first administration of IMP. History or evidence of any other clinically significant disorder (eg, cognitive impairment), condition or disease other than those outlined above that, in the opinion of the Investigator or AstraZeneca physician, if consulted, may compromise the ability of the subject to give written informed consent, would pose a risk to subject safety, or interfere with the study evaluation, procedures or completion.

33. Subject likely to not be available to complete all protocol required study visits or procedures, to the best of the subject's and Investigator's knowledge.

34. Non-leukocyte depleted whole blood transfusion within 120 days of the date of the genetic sample collection.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2019-11-21 (Actual); Primary Completion 2021-06-07 (Actual); Study Completion 2021-06-07 (Actual)

PRIMARY OUTCOMES:
Number of subjects with adverse events (AEs) due to AZD8233 SC multiple ascending dose treatment. | From randomization to final Follow-up Visit (Week 16 post last dose).
  To assess AEs as a variable of safety and tolerability of AZD8233 following SC administration of multiple ascending doses. Serious AEs will be recorded from the time of informed consent.
Vital sign: Systolic blood pressure (SBP) | From screening to final Follow-up Visit (Week 16 post last dose).
  To assess SBP as a variable of safety and tolerability of AZD8233 following SC administration of multiple ascending doses. BP will be collected after the subject has rested in the supine position for at least 5 minutes.
Vital sign: Pulse rate | From screening visit to final Follow-up Visit (Week 16 post last dose).
  To assess supine position pulse as a variable of safety and tolerability of AZD8233 following SC administration of multiple ascending doses. Pulse rate will be collected after the subject has rested in the supine position for at least 5 minutes.
Vital sign: Oral body temperature | Day -1 to final Follow-up Visit (Week 16 post last dose).
  To assess the oral body temperature as a variable of safety and tolerability of AZD8233 following SC administration of multiple ascending doses.
Number of patients with abnormal findings in resting 12-lead Electrocardiogram (ECG) and digital ECG (dECG). | From screening to final Follow-up Visit (Week 16 post last dose).
  To assess the clinically significant abnormalities in the cardiovascular system functioning using a 12-lead ECG as a variable of safety and tolerability of AZD8233 following SC administration of multiple ascending doses. ECG evaluations will be recorded after approximately 10 min resting in supine position. dECGs will be done only on Days 1 and 57 (pre-dose and at 0.5, 1, 2, 3, 4, 6, 8, 12 and 24, 36 and 48 hours post-dose), and Days 8 and 29 (pre-dose).
Number of subject with abnormal findings in cardiac telemetry | At Day -1, Days 1 to 3 (pre-dose to 24 hours post-dose), and Day 57 (pre-dose to 24 hours post-dose).
  To assess cardiac telemetry as a variable of safety and tolerability of AZD8233 following SC administration of multiple ascending doses.
Physical examination | From screening to final Follow-up Visit (Week 16 post last dose).
  To assess physical examination as a variable of safety and tolerability of AZD8233 following SC administration of multiple ascending doses. Complete (general appearance, respiratory, cardiovascular, abdomen, skin, head and neck [including ears, eyes, nose and throat], lymph nodes, thyroid, musculoskeletal [including spine and extremities] and neurological systems).
Injection site reaction examinations | From randomization to final Follow-up Visit (Week 16 post last dose).
  To assess injection site reactions in terms of size (mm), color (pale/light red/dark red), and itching (yes or no)as a variable of safety and tolerability of AZD8233 following SC administration of multiple ascending doses.
Laboratory assessments: Hematology - Blood cells count | From screening to final Follow-up Visit (Week 16 post last dose).
  To assess red blood cells (RBC) and white blood cells (WBC) as a variable of safety and tolerability of AZD8233 following SC administration of multiple ascending doses.
Laboratory assessments: Hematology - Hemoglobin (Hb) | From screening to final Follow-up Visit (Week 16 post last dose).
  To assess Hb as a variable of safety and tolerability of AZD8233 following SC administration of multiple ascending doses.
Laboratory assessments: Hematology - Hematocrit (HCT) | From screening to final Follow-up Visit (Week 16 post last dose).
  To assess HCT as a variable of safety and tolerability of AZD8233 following SC administration of multiple ascending doses.
Laboratory assessments: Hematology - Mean corpuscular volume (MCV) | From screening to final Follow-up Visit (Week 16 post last dose).
  To assess MCV as a variable of safety and tolerability of AZD8233 following SC administration of multiple ascending doses.
Laboratory assessments: Hematology - Mean corpuscular hemoglobin (MCH) | From screening to final Follow-up Visit (Week 16 post last dose).
  To assess MCH as a variable of safety and tolerability of AZD8233 following SC administration of multiple ascending doses.
Laboratory assessments: Hematology - Mean corpuscular hemoglobin concentration (MCHC) | From screening to final Follow-up Visit (Week 16 post last dose).
  To assess MCHC as a variable of safety and tolerability of AZD8233 following SC administration of multiple ascending doses.
Laboratory assessments: Hematology - Differential WBC count | From screening to final Follow-up Visit (Week 16 post last dose).
  To assess differential WBC count absolute count of neutrophils, lymphocytes, monocytes, eosinophils and basophils as a variable of safety and tolerability of AZD8233 following SC administration of multiple ascending doses.
Laboratory assessments: Hematology - Platelet count and platelet function assessment. | From screening to final Follow-up Visit (Week 16 post last dose).
  To assess platelet count and platelet function in platelet rich plasma (PRP) using Light Transmission Aggregometry (LTA) as a variable of safety and tolerability of AZD8233 following SC administration of multiple ascending doses.
Laboratory assessments: Hematology - Reticulocytes absolute count | From screening to final Follow-up Visit (Week 16 post last dose).
  To assess Reticulocytes absolute count as a variable of safety and tolerability of AZD8233 following SC administration of multiple ascending doses.
Laboratory assessments: Serum clinical chemistry - Electrolytes | From screening to final Follow-up Visit (Week 16 post last dose).
  To assess serum level of sodium, potassium, calcium as a variable of safety and tolerability of AZD8233 following SC administration of multiple ascending doses.
Laboratory assessments: Serum clinical chemistry - Blood urea nitrogen (BUN) | From screening to final Follow-up Visit (Week 16 post last dose).
  To assess serum level of BUN as a variable of safety and tolerability of AZD8233 following SC administration of multiple ascending doses.
Laboratory assessments: Serum clinical chemistry - Creatinine | From screening to final Follow-up Visit (Week 16 post last dose).
  To assess serum level of creatinine as a variable of safety and tolerability of AZD8233 following SC administration of multiple ascending doses.
Laboratory assessments: Serum clinical chemistry - Glucose (fasting) | From screening to final Follow-up Visit (Week 16 post last dose).
  To assess serum fasting glucose level as a variable of safety and tolerability of AZD8233 following SC administration of multiple ascending doses.
Laboratory assessments: Serum clinical chemistry - Creatine kinase | From screening to final Follow-up Visit (Week 16 post last dose).
  To assess the level of serum creatine kinase as a variable of safety and tolerability of AZD8233 following SC administration of multiple ascending doses.
Laboratory assessments: Serum clinical chemistry - Direct bilirubin | From screening to final Follow-up Visit (Week 16 post last dose).
  To assess the level of serum bilirubin (direct) as a variable of safety and tolerability of AZD8233 following SC administration of multiple ascending doses.
Laboratory assessments: Serum clinical chemistry - Hemoglobin A1c (HbA1c) | From screening to final Follow-up Visit (Week 16 post last dose).
  To assess the level of HbA1c as a variable of safety and tolerability of AZD8233 following SC administration of multiple ascending doses.
Laboratory assessments: Serum clinical chemistry - Liver enzymes | From screening to final Follow-up Visit (Week 16 post last dose).
  To assess the level of Alkaline phosphatase (ALP), Alanine aminotransferase (ALT), Aspartate aminotransferase (AST), and Gamma glutamyl transpeptidase (GGT) as a variable of safety and tolerability of AZD8233 following SC administration of multiple ascending doses.
Laboratory assessments: Serum clinical chemistry - Total bilirubin | From screening to final Follow-up Visit (Week 16 post last dose).
  To assess the level of serum bilirubin (total) as a variable of safety and tolerability of AZD8233 following SC administration of multiple ascending doses.
Laboratory assessments: Serum clinical chemistry - Cell enzymes | From screening to final Follow-up Visit (Week 16 post last dose).
  To assess the level of serum glutamate dehydrogenase (GLDH) and lactate dehydrogenase (LDH) as a variable of safety and tolerability of AZD8233 following SC administration of multiple ascending doses.
Laboratory assessments: Serum clinical chemistry - Bicarbonate | From screening to final Follow-up Visit (Week 16 post last dose).
  To assess the level of bicarbonate as a variable of safety and tolerability of AZD8233 following SC administration of multiple ascending doses.
Laboratory assessments: Serum clinical chemistry - Uric acid | From screening to final Follow-up Visit (Week 16 post last dose).
  To assess the level of uric acid as a variable of safety and tolerability of AZD8233 following SC administration of multiple ascending doses.
Laboratory assessments: Coagulation | From screening to final Follow-up Visit (Week 16 post last dose).
  To assess activated partial thrombin time (aPTT), prothrombin time (PT), and International normalized ratio (INR) as a variable of safety and tolerability of AZD8233 following SC administration of multiple ascending doses.
Renal safety biomarkers - Urine clusterin | Screening, Day 1 (pre-dose, 24 hours and 48 hours post-dose), Days 8 and 29 (pre-dose), and Day 57 (pre-dose).
  To assess renal biomarker by evaluation of urine clusterin level as a variable of safety and tolerability of AZD8233 following SC administration of multiple ascending doses.
Renal safety biomarkers - Urine cystatin-C | Screening, Day 1 (pre-dose, 24 hours and 48 hours post-dose), Days 8 and 29 (pre-dose), and Day 57 (pre-dose).
  To assess renal biomarker by evaluation of urine cystatin-C level as a variable of safety and tolerability of AZD8233 following SC administration of multiple ascending doses.
Renal safety biomarkers - Urine N-acetyl-beta-D-glucosaminidase (NAG) | Screening, Day 1 (pre-dose, 24 hours and 48 hours post-dose), Days 8 and 29 (pre-dose), and Day 57 (pre-dose).
  To assess renal biomarker by evaluation of urine NAG level as a variable of safety and tolerability of AZD8233 following SC administration of multiple ascending doses.
Renal safety biomarkers - Urine albumin | Screening, Day 1 (pre-dose, 24 hours and 48 hours post-dose), Days 8 and 29 (pre-dose), and Day 57 (pre-dose).
  To assess renal biomarker by evaluation of urine albumin level as a variable of safety and tolerability of AZD8233 following SC administration of multiple ascending doses.
Renal safety biomarkers - Urine creatinine | Screening, Day 1 (pre-dose, 24 hours and 48 hours post-dose), Days 8 and 29 (pre-dose), and Day 57 (pre-dose).
  To assess renal biomarker by evaluation of urine creatinine level as a variable of safety and tolerability of AZD8233 following SC administration of multiple ascending doses.
Renal safety biomarkers - Urine Kidney injury molecule1 (KIM-1) | Screening, Day 1 (pre-dose, 24 hours and 48 hours post-dose), Days 8 and 29 (pre-dose), and Day 57 (pre-dose).
  To assess renal biomarker by evaluation of urine KIM-1 level as a variable of safety and tolerability of AZD8233 following SC administration of multiple ascending doses.
Renal safety biomarkers - Urine Neutrophil gelatinase-associated lipocalin (NGAL) | Screening, Day 1 (pre-dose, 24 hours and 48 hours post-dose), Days 8 and 29 (pre-dose), and Day 57 (pre-dose).
  To assess renal biomarker by evaluation of urine NAG level as a variable of safety and tolerability of AZD8233 following SC administration of multiple ascending doses.
Renal safety biomarkers - Urine Osteopontin | Screening, Day 1 (pre-dose, 24 hours and 48 hours post-dose), Days 8 and 29 (pre-dose), and Day 57 (pre-dose).
  To assess renal biomarker by evaluation of urine osteopontin level as a variable of safety and tolerability of AZD8233 following SC administration of multiple ascending doses.
Renal safety biomarkers - Urine total protein | Screening, Day 1 (pre-dose, 24 hours and 48 hours post-dose), Days 8 and 29 (pre-dose), and Day 57 (pre-dose).
  To assess renal biomarker by evaluation of urine protein (total) level as a variable of safety and tolerability of AZD8233 following SC administration of multiple ascending doses.
Immune Activation Response - High-sensitivity C-reactive protein (hs-CRP) | From screening to final Follow-up Visit (Week 16 post last dose).
  To assess hs-CRP level as a variable of safety and tolerability of AZD8233 following SC administration of multiple ascending doses.
Complement Activation panel | Days 1 and 57 (pre-dose, 1, 2, and 4 hours post-dose).
  To assess chemotactic factor (C3a, Bb, and C5a) levels as a variable of safety and tolerability of AZD8233 following SC administration of multiple ascending doses.
Laboratory assessments: Clinical urinalysis | From screening to final Follow-up Visit (Week 16 post last dose).
  To assess urine sample for proteins, blood, creatinine, microscopy evaluation as a variable of safety and tolerability of AZD8233 following SC administration of multiple ascending doses.

SECONDARY OUTCOMES:
Plasma PK analysis: Time delay between drug administration and the first observed concentration in plasma (tlag). | Days 1 and 57 (Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48 hours post-dose); Day 8 (pre-dose), Days 15, 22, 29 (pre-dose), Days 36 and 44.
  To characterize the tlag of AZD8233 following SC administration of multiple ascending doses.
Plasma PK analysis: Time to reach peak or maximum observed concentration or response following drug administration (tmax). | Days 1 and 57 (Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48 hours post-dose); Day 8 (pre-dose), Days 15, 22, 29 (pre-dose), Days 36 and 44.
  To characterize the tmax of AZD8233 following SC administration of multiple ascending doses.
Plasma PK analysis: Observed maximum plasma concentration (Cmax). | Days 1 and 57 (Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48 hours post-dose); Day 8 (pre-dose), Days 15, 22, 29 (pre-dose), Days 36 and 44.
  To characterize the Cmax of AZD8233 following SC administration of multiple ascending doses.
Plasma PK analysis: Area under the plasma concentration-curve from time zero to time last value above the limit of quantification (AUC[0-last]). | Days 1 and 57 (Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48 hours post-dose); Day 8 (pre-dose), Days 15, 22, 29 (pre-dose), Days 36 and 44.
  To characterize the AUC(0-last) of AZD8233 following SC administration of multiple ascending doses.
Plasma PK analysis: Area under the concentration-time curve from time zero to 24 hours post-dose (AUC[0-24]). | Days 1 and 57 (Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48 hours post-dose); Day 8 (pre-dose), Days 15, 22, 29 (pre-dose), Days 36 and 44.
  To characterize the AUC(0-24) of AZD8233 following SC administration of multiple ascending doses.
Plasma PK analysis: Area under the concentration-time curve from time zero to 48 hours post-dose (AUC[0-48]). | Days 1 and 57 (Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48 hours post-dose); Day 8 (pre-dose), Days 15, 22, 29 (pre-dose), Days 36 and 44.
  To characterize the AUC(0-48) of AZD8233 following SC administration of multiple ascending doses.
Plasma PK analysis: Area under the concentration-time curve from time zero extrapolated to infinity (AUC). | Days 1 and 57 (Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48 hours post-dose); Day 8 (pre-dose), Days 15, 22, 29 (pre-dose), Days 36 and 44.
  To characterize the AUC of AZD8233 following SC administration of multiple ascending doses. AUC is estimated by AUC(0-last) + Clast/λz where Clast is the last observed quantifiable concentration.
Plasma PK analysis: Area under the plasma concentration-time curve from time during the dosing interval (AUCt). | Days 1 and 57 (Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48 hours post-dose); Day 8 (pre-dose), Days 15, 22, 29 (pre-dose), Days 36 and 44.
  To characterize the AUCt of AZD8233 following SC administration of multiple ascending doses.
Plasma PK analysis: Observed trough plasma drug concentration (Ctrough). | Days 1 and 57 (Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48 hours post-dose); Day 8 (pre-dose), Days 15, 22, 29 (pre-dose), Days 36 and 44.
  To characterize the Ctrough of AZD8233 following SC administration of multiple ascending doses.
Plasma PK analysis: Apparent total body clearance of drug from plasma after extravascular administration (CL/F). | Days 1 and 57 (Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48 hours post-dose); Day 8 (pre-dose), Days 15, 22, 29 (pre-dose), Days 36 and 44.
  To characterize the CL/F of AZD8233 following SC administration of multiple ascending doses.
Plasma PK analysis: Apparent volume of distribution for parent drug at terminal phase (extravascular administration) (Vz/F). | Days 1 and 57 (Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48 hours post-dose); Day 8 (pre-dose), Days 15, 22, 29 (pre-dose), Days 36 and 44.
  To characterize the Vz/F of AZD8233 following SC administration of multiple ascending doses; estimated by dividing the apparent clearance (CL/F) by λz.
Plasma PK analysis: Half-life associated with the terminal slope (λz) of a semi-logarithmic concentration-time curve (t1/2). | Days 1 and 57 (Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48 hours post-dose); Day 8 (pre-dose), Days 15, 22, 29 (pre-dose), Days 36 and 44.
  To characterize the t1/2 of AZD8233 following SC administration of multiple ascending doses.
Plasma PK analysis: Mean Residence Time (MRT). | Days 1 and 57 (Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48 hours post-dose); Day 8 (pre-dose), Days 15, 22, 29 (pre-dose), Days 36 and 44.
  To characterize the MRT of AZD8233 following SC administration of multiple ascending doses.
Urine PK analysis: Amount excreted in urine (Ae). | Treatment Days 1 to 3 (Pre-dose and intervals 0-6, 6-12 hours and 12-24 hours post-dose).
  To characterize the Ae of AZD8233 following SC administration of multiple ascending doses.
Urine PK analysis: Fraction excreted unchanged in urine (Fe). | Treatment Days 1 to 3 (Pre-dose and intervals 0-6, 6-12 hours and 12-24 hours post-dose).
  To characterize the Fe of AZD8233 following SC administration of multiple ascending doses.
Urine PK analysis: Renal clearance (CLR). | Treatment Days 1 to 3 (Pre-dose and intervals 0-6, 6-12 hours and 12-24 hours post-dose).
  To characterize the CLR of AZD8233 following SC administration of multiple ascending doses.
PD analysis: Levels of dyslipidemia related biomarkers. | At screening, Day -1, Days 1 to 3 and Days 57 to 58 (pre-dose and 48 hours post-dose), Day 8 (pre-dose), Days 15, 22, Day 29 (pre-dose), Days 36, 44, Day 56, week 2 to 14 (at 2, 4, 6, 8, 10, 12, and 14 weeks) and week 16 post-dose.
  To assess the effect of AZD8233 on levels of dyslipidemia related biomarkers.

CONTACTS AND LOCATIONS:
Overall Officials: David Han, MD, Principal Investigator — PAREXEL Early Phase Clinical Unit-Los Angeles
Locations (7):
- United States (7):
  - Research Site, Chula Vista, California
  - Research Site, Glendale, California
  - Research Site, La Mesa, California
  - Research Site, Jacksonville, Florida
  - Research Site, Orlando, Florida
  - Research Site, Port Orange, Florida
  - Research Site, Brooklyn, Maryland

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the European Federation of Pharmaceutical Industries and Associations Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Clewe O, Rekic D, Quartino AL, Carlsson B, Higashimori M, Wernevik L, Hofherr A, Ryden-Bergsten T, Nilsson C, Knochel J. Population pharmacokinetics of a novel PCSK9 antisense oligonucleotide. Br J Clin Pharmacol. 2024 Jun;90(6):1503-1513. doi: 10.1111/bcp.16046. Epub 2024 Mar 19. PMID 38504437